CLINICAL TRIAL: NCT03557177
Title: Clinical Characterisation of the Vascular Effects of Cis-platinum Based Chemotherapy in Patients With Testicular Cancer
Acronym: VECTOR
Status: Completed | Type: Observational
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Sponsor
Other Study IDs: GN15CA467
Record Dates: First submitted 2018-06-04; First posted 2018-06-14 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Testicular Cancer; Cardiovascular Diseases
Keywords: cisplatin; flow mediated dilatation
MeSH Terms: conditions — Testicular Neoplasms; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biological blood samples will be retained without DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
incidence is increasing1,2. Whilst the prognosis is very good with the vast majority of patients cured with orchidectomy alone, those with high risk stage one non seminomatous germ cell cancer (NSCGT) or metastatic disease (NSCGT or seminoma) are treated by surgery followed by chemotherapy. Platinum based chemotherapy is associated with long-term cardiovascular sequelae.

Endothelial dysfunction is a key component of early atherogenesis and the later stages of obstructive atherosclerosis, plaque rupture and thrombus formation. Whilst endothelial toxic effects of BEP chemotherapy appear to be central in the pathophysiology of associated complications, abnormalities in endothelial function as assessed by measures of brachial artery flow-mediated dilatation (FMD) have not demonstrated a consistent effect over time. When assessed within ten weeks of platinum-based chemotherapy9, no change in FMD was observed whilst marked decreases are seen immediately following treatment11 and also one year following treatment12. Therefore, the time-course of endothelial vasomotor impairment remains incompletely defined in a single prospective cohort.

DETAILED DESCRIPTION:
There remains an unmet need to identify a preventive treatment for patients with testicular cancer treated with platinum based chemotherapy to diminish the substantial risk of subsequent cardiovascular events. A future randomised trial of statin therapy in these patients is under consideration and results from this pilot study will inform its design.

Before moving towards interventional studies the proposed pilot study will enable a better understanding of the nature, time-course and dose-dependent effects of the mechanisms contributing to increased cardiovascular risk.

Single-centre, prospective pilot study assessing the cardiovascular effects of treatment with orchidectomy or orchidectomy plus cisplatin based chemotherapy for testicular cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of stage 1 or IGCCCG5good or intermediate prognosis metastatic testicular/retroperitoneal germ cell cancer with treatment plan that includes orchidectomy or orchidectomy plus cisplatin based chemotherapy
* Aged between 18 and 65 years inclusive

Exclusion Criteria:

* Unable to provide written, informed consent
* Unable or unwilling to attend for investigations
* Current involvement in a clinical trial
* Anti-platelet therapy at time of enrolment
* Statin or other lipid-lowering therapy at time of enrolment
* Recreational drug use
* Ongoing inflammatory, infective or autoimmune disease
* Other malignant disease diagnosed in previous 5 years
* Previous venous or arterial thrombotic/thromboembolic event

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orchidectomy alone or Orchidectomy plus 1-2 cycles adjuvant cisplatin based chemotherapy or Orchidectomy plus 3-4 cycles cisplatin based chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Change in flow-mediated dilatation post cisplatin based chemotherapy | 9 months
  Maximum change in flow-mediated dilatation post cisplatin based chemotherapy

SECONDARY OUTCOMES:
Percentage change in circulating platelet monocyte aggregates post cisplatin based chemotherapy | 9 months
  Maximum change in percentage circulating platelet monocyte aggregates post cisplatin based chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Ninian Lang, MBChB PhD, Principal Investigator — QEUH, NHS Greater Glasgow and Clyde
Locations (1):
- Beatson West of Scotland Cancer Centre, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided